CLINICAL TRIAL: NCT03069820
Title: Clarify of Predictive Risk Factors of Chemotherapy-induced Liver Injury After Therapy With Docetaxel and Cisplatin for Nasopharyngeal Carcinoma
Brief Title: Clarify of Predictive Risk Factors of Chemotherapy-induced Liver Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HL001
Record Dates: First submitted 2017-02-13; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Liver Injury, Drug-Induced
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): Patients with advanced nasopharyngeal carcinoma scheduled to receive the first line, first cycle TP (docetaxel and cisplatin) chemotherapy
  Interventions: Drug: docetaxel and cisplatin

INTERVENTIONS:
Drug: docetaxel and cisplatin — Patients receive TP (docetaxel and cisplatin) chemotherapy
  Other Names: Taxotere

SUMMARY:
The most common toxicity of TP (docetaxel and cisplatin) chemotherapy is chemotherapy-induced liver injury. However, patients don't always experience same chemotherapy-induced liver injury for the same drugs. Therefore, the investigators designed the present study to clarify risk factors associated with the development of severe hepatotoxicity after therapy with docetaxel and cisplatin for nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignancies in southern China , with an annual incidence of 15 to 50 cases per 100,000 people. NPC is both radiosensitive and chemosensitive. Recently, many new drugs including docetaxel and cisplatin have been incorporated in the induction chemotherapy phase of NPC. The most common toxicity of TP (docetaxel and cisplatin) chemotherapy is chemotherapy-induced liver injury, and appropriate management of these toxicities can help patients improve tolerance for chemotherapy. However, patients don't always experience same chemotherapy-induced liver injury for the same drugs. Therefore, it is important to determine the risk factors to predict chemotherapy-induced liver injury. The investigators designed the present study to clarify risk factors associated with the development of severe hepatotoxicity after therapy with docetaxel and cisplatin for nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced nasopharyngeal carcinoma.
* Patients scheduled to receive the first line, first cycle TP (docetaxel and cisplatin) chemotherapy.
* Normal liver function biomarkers including ALT,AST,ALP,TBIL before recruitment.
* Minimum age of 18 years.
* Life expectancy at least 3 months.

Exclusion Criteria:

* Patients previously received chemotherapy
* Patients who have liver metastases.
* Patients who take other drugs that may affect liver function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Relationship of white blood cell level and chemotherapy-induced liver injury | 3 weeks
  White blood cell level (cells/L) and liver function (such as ALT, AST, ALP, and bilirubin levels) will be tested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy, and the relationship of white cell level fluctuation and liver injury will be investigated.
Relationship of albumin level and chemotherapy-induced liver injury | 3 weeks
  Albumin (g/L) and liver function (such as ALT, AST, ALP, and bilirubin levels) will be tested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy, and the relationship of albumin fluctuation and liver injury will be investigated.
Relationship of hemoglobin level and chemotherapy-induced liver injury | 3 weeks
  Hemoglobin (g/L) and liver function (such as ALT, AST, ALP, and bilirubin levels) will be tested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy, and the relationship of hemoglobin fluctuation and liver injury will be investigated.
Relationship of blood platelet level and chemotherapy-induced liver injury | 3 weeks
  Blood platelet (cells/L) and liver function (such as ALT, AST, ALP, and bilirubin levels) will be tested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy, and the relationship of blood platelet fluctuation and liver injury will be investigated.

SECONDARY OUTCOMES:
Relationship of age and chemotherapy-induced liver injury | 3 weeks
  The age(years) will be recorded when the therapy starts. The liver function (such as ALT, AST, ALP, and bilirubin levels) will betested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy. The relationship of age and liver injury will be investigated.
Relationship of height and chemotherapy-induced liver injury | 3 weeks
  The height (kg) will be recorded when the therapy starts. The liver function (such as ALT, AST, ALP, and bilirubin levels) will betested before (1-3 days) and after (21 ± 3 days) first cycle of chemotherapy. The relationship of height and liver injury will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Long Huang, MD, Study Director — The Second Afiliated Hospital of Nanchang University
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No